CLINICAL TRIAL: NCT01355354
Title: An Open-Label, Non-Randomised, 2-Period, Single Centre Study to Assess the Pharmacokinetics of Digoxin in Healthy Subjects When Administered Alone and in Combination With Fostamatinib 100 mg Twice Daily
Brief Title: Effects of Administration of Fostamatinib on Blood Concentrations of Digoxin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D4300C00026
Record Dates: First submitted 2011-05-17; First posted 2011-05-18 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Healthy Volunteers; Rheumatoid Arthritis
Keywords: Phase 1; healthy volunteers; pharmacokinetics; Rheumatoid arthritis; RA, Fostamatinib; Digoxin, drug-drug interaction; Scientific terminology: Rheumatoid arthritis; Fostamatinib; Digoxin; drug-drug interaction; Laymen terminology: Rheumatoid arthritis; Amount of Digoxin in blood
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Digoxin; fostamatinib

ARMS (2):
- 1 (Experimental): Digoxin
  Interventions: Drug: Digoxin
- 2 (Experimental): Fostamatinib
  Interventions: Drug: Digoxin; Drug: Fostamatinib

INTERVENTIONS:
Drug: Digoxin — oral tablets, 0.25mg bd on Day 1 and 0.25 Once daily from Day 2 to 15
Drug: Fostamatinib — oral tablets, 100mg (2 X 50mg) bd from Day 9 - 15
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the drug interaction between fostamatinib and digoxin by comparing the safety, tolerability and plasma concentration of digoxin when administered alone and with fostamatinib in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Male or female subjects aged 18 to 45 years (inclusive)
* Minimum weight of 50 kg and body mass index (BMI) between 18 and 30 kg/m2 (inclusive)
* Female subjects must have a negative pregnancy test at screening and on Day -1,must not be lactating, and must be of non-childbearing potential

Exclusion Criteria:

* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs (except for cholecystectomy)
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of the investigational product
* Subjects who smoke more than 5 cigarettes or the equivalent in tobacco per day
* Absolute neutrophil count of <2500/mm3 or 2.5 x 109/L
* Previous treatment with fostamatinib or digoxin in the present study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To investigate whether the plasma concentration-time profiles and resulting PK parameters of digoxin are altered during steady-state fostamatinib administration. Digoxin AUCss and Cmaxss will be measured | Day 8 and Day 15

SECONDARY OUTCOMES:
To examine the safety + tolerability of fostamatinib in combination with digoxin. Assessments: Adverse events, lab assessments, vital signs, phys exam,12-lead ECG. Absolute values and change in baseline for any of these parameters will be reported | From screening, Day 1 - Day 17, through to Follow up visit
To examine the steady-state PK of R406 during co-administration of fostamatinib with digoxin at steady-state. R406 AUCss, tmaxss and Cmaxss will be measured | Day 15
To examine the urinary steady-state PK of digoxin in healthy subjects when administered alone and in combination with fostamatinib at steady-state. Digoxin Ae(0-t), Fe, and CLr will be measured | Day 8 and Day 15

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- [Derived] Martin P, Gillen M, Millson D, Oliver S, Brealey C, Elsby R, Baluom M, Lau D, Mant T. Effects of Fostamatinib on the Pharmacokinetics of Digoxin (a P-Glycoprotein Substrate): Results From in Vitro and Phase I Clinical Studies. Clin Ther. 2015 Dec 1;37(12):2811-22. doi: 10.1016/j.clinthera.2015.09.018. Epub 2015 Oct 26. PMID 26514315